# **Study Protocol**

## **Official Title:**

Effectiveness of a Multimodal Information Technology-enhanced Hand Hygiene Improvement Strategy on Healthcare-associated Infections in Nursing Homes

**NCT Number**:

NCT06925620

**Document Date:** 

January 27, 2022

### **Study Protocol**

### **Study Objectives:**

- 1. To evaluate the effect of a multimodal hand hygiene intervention on healthcare workers' hand hygiene knowledge, compliance, and technique accuracy.
- 2. To assess the impact of the intervention on healthcare-associated infection (HAI) density rates in nursing homes.

## **Study Design:**

- 1. Cluster-randomized controlled trial.
- 2. Four nursing homes were randomly assigned to the experimental group (two facilities) or the control group (two facilities).

#### **Participants:**

- 1. Nurses and nursing assistants working in participating nursing homes.
- 2. Inclusion: Currently employed staff.
- 3. Exclusion: Individuals who had submitted their resignation.

#### **Intervention:**

- 1. Experimental group: Received a three-month multimodal IT-enhanced hand hygiene program including amenities, reminders, education, observation with feedback, and patient safety climate improvements.
- 2. Control group: Continued routine hand hygiene practices.

#### **Outcome Measures:**

- 1. Primary outcome: Hand hygiene knowledge, technique accuracy, and compliance.
- 2. Secondary outcome: Healthcare-associated infection density.

**Data Collection**: Baseline and post-intervention at 1, 2, and 3 months.

**Ethical Approval**: Approved by Kaohsiung Medical University Chung-Ho Memorial Hospital Institutional Review Board (KMUHIRB-F(I)-20220007).

**Confidentiality**: Participant data will be anonymized and securely stored.

**Publication Policy**: Results will be published in journals.